CLINICAL TRIAL: NCT05583526
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, 52-WEEK PLACEBO-CONTROLLED, MULTI-CENTER STUDY INVESTIGATING THE EFFICACY, SAFETY, AND TOLERABILITY OF RITLECITINIB IN ADULT AND ADOLESCENT PARTICIPANTS WITH NON SEGMENTAL VITILIGO
Brief Title: A 52-Week Study of Ritlecitinib Oral Capsules in Adults and Adolescents With Nonsegmental Vitiligo (Active and Stable) Tranquillo
Acronym: Tranquillo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981040; Tranquillo (Other: Alias Study Number); 2022-501668-16-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-06; First posted 2022-10-17 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Stable Nonsegmental Vitiligo; Active Nonsegmental Vitiligo

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel-group, vehicle controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ritlecitinib 50 mg (Experimental): Ritlecitinib 50 mg QD (ritilecitinib 50 mg QD arm; approximately 400 participants)
  Interventions: Drug: Ritlecitinib
- Placebo (Placebo Comparator): Placebo (placebo arm; approximately 200 participants)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ritlecitinib — 50 mg capsule
  Arms: Ritlecitinib 50 mg
Drug: Placebo — Matching capsule
  Arms: Placebo

SUMMARY:
A 52-Week Study of Ritlecitinib Oral Capsules in Adults and Adolescents with Nonsegmental Vitiligo (Active and Stable) Tranquillo

DETAILED DESCRIPTION:
Study B7981040 is a Phase 3 randomized, double-blind, 52-week placebo-controlled, multi center study investigating the efficacy, safety, and tolerability of ritlecitinib in adult and adolescent participants with nonsegmental vitiligo (both active and stable vitiligo).

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years of age at Screening. Adolescents (12 to <18 years of age) are also eligible for this study, but only if approved by the local IRB/EC and regulatory health authority. Where these approvals have not been granted, only participants ≥18 years of age will be enrolled.

   Disease Characteristics:
2. Eligible participants must have at both Screening and Baseline:

   * A clinical diagnosis of nonsegmental vitiligo for at least 3 months; and
   * BSA involvement 4%-60% inclusive, excluding involvements at palms of the hands, soles of the feet, or dorsal aspect of the feet; and
   * BSA ≥0.5% involvement on the face (face is defined as including the area on the forehead to the original hairline, on the cheek vertically to the jawline, and laterally from the corner of the mouth to the tragus. The face will not include scalp, ears, neck, or surface area of the lips, but will include the nose and the eyelids; and
   * F-VASI ≥0.5 & T-VASI ≥3; and
   * Either active or stable disease nonsegmental vitiligo at both Screening and Baseline visits. All participants who do not have the features of active vitiligo (defined below) are required to have stable disease.

   Active vitiligo is defined as:
   * Participants will be classified as having active vitiligo based on the presence of at least one active lesion at baseline defined as one of the following:
   * New/extending lesion(s) in the 3 months prior to Screening visit (confirmed by photographs or medical record):
   * Confetti-like lesion(s); Confetti-like depigmentation is characterized by the presence of numerous 1-mm to 5-mm depigmented macules in clusters;
   * Trichrome lesion(s);Trichrome lesions have a hypopigmented zone of varying width between normal and completely depigmented skin, resulting in 3 different hues of skin;
   * Koebner phenomenon/phenomena (excluding Type 1 [history based on isomorphic reaction]). The Koebner phenomenon manifests as depigmentation at sites of trauma, usually in a linear arrangement.

   Stable vitiligo is defined as an absence of signs of active disease. All participants who do not have the features of active vitiligo (defined above) are required to have stable disease.

   Eligibility is determined at Screening and Baseline based on the resulting scores from the local in-person reads of F-VASI, T-VASI, and BSA.

   Other Inclusion Criteria:
3. If receiving concomitant medications for any reason other than vitiligo, participant must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1. Participant must be willing to stay on a stable regimen during the duration of the study.
4. Must agree to stop all other treatments for vitiligo from Screening through the final follow-up visit.

Exclusion Criteria:

1. Any psychiatric condition including recent or active suicidal ideation or behavior that meets any of the following criteria:

   * Suicidal ideation associated with actual intent and a method or plan in the past year: "Yes" answers on items 4 or 5 of the C-SSRS administered at the screening visit.
   * Previous history of suicidal behaviors in the past 5 years: "Yes" answer (for events that occurred in the past 5 years) to any of the suicidal behavior items of the C-SSRS.
   * For adults, any lifetime history of serious suicidal behavior or recurrent suicidal behavior. For adolescents, any previous lifetime history of suicidal behavior.
2. Medical conditions pertaining to vitiligo and other diseases/conditions affecting the skin:

   * Participants that have other types of vitiligo that do not meet criteria for active or stable vitiligo as noted in inclusion criterion #2 (including, but not limited to, segmental vitiligo and mixed vitiligo).
   * Currently have active forms of other disorders of pigmentation (including but not limited to Vogt-Koyanagi-Harada disease, malignancy-induced hypopigmentation [melanoma and mycosis fungoides], post-inflammatory hypopigmentation, pityriasis alba [minor manifestation of atopic dermatitis], senile leukoderma [age-related depigmentation], chemical/drug-induced leukoderma, ataxia telangiectasia, tuberous sclerosis, melasma (all types, including mixed), and congenital hypopigmentation disorder including piebaldism, Waardenburg syndrome, hypomelanosis of Ito, incontinentia pigmenti, dyschromatosis symmetrica hereditarian, xeroderma pigmentosum, and nevus depigmentosus). NOTE: Coexistence of halo nevus/nevi (also known as Sutton nevus/nevi) is permitted.
   * Currently have active forms of inflammatory skin disease(s) or evidence of skin conditions (for example, morphea, discoid lupus, leprosy, syphilis, psoriasis, seborrheic dermatitis) at the time of the Screening or Baseline Visit that in the opinion of the investigator would interfere with evaluation of vitiligo or response to treatment.
   * Leukotrichia in more than 33% of the face surface area affected with vitiligo lesions OR leukotrichia in more than 33% of the total body surface area affected with vitiligo lesions.
   * Have a superficial skin infections within 2 weeks prior to first dose on Day 1. NOTE: participants may be rescreened after the infection resolves.
3. General Infection History:

   * Having a history of systemic infection requiring hospitalization, parenteral antimicrobial, antiviral (including biologic treatment), antiparasitic, antiprotozoal, or antifungal therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1.
   * Have active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 1. NOTE: participants may be rescreened after the infection resolves.
   * Evidence or history of untreated, currently treated or inadequately treated active or latent infection with Mycobacterium TB
4. Specific Viral Infection History:

   * History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
   * Infected with hepatitis B or hepatitis C viruses: all participants will undergo screening for hepatitis B and C for eligibility.
   * Participants who are positive for HCVAb and HCV RNA will not be eligible for this study.
   * Have a known immunodeficiency disorder (including positive serology for HIV at screening) or a first-degree relative with a hereditary immunodeficiency.
5. Medical Conditions, Other:

   * Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (eg, untreated hypovitaminosis D or hypothyroidism), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator or Pfizer (or designee), the participant is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle requirements.
   * History of severe allergic or anaphylactoid reaction to any kinase inhibitor or a known allergy/hypersensitivity to any component (including excipients) of the study intervention.
   * Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating or progressive.
   * Have a history of any lymphoproliferative disorder such as EBV-related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
   * Abnormal findings on the Screening chest imaging (eg, chest x-ray) that may increase the risk associated with study participation including, but not limited to, presence of active TB, general infections, cardiomyopathy, or malignancy. Chest imaging may be performed up to 12 weeks prior to screening. Documentation of the official reading must be located and available in the source documentation.
   * Long QT Syndrome, a family history of Long QT Syndrome, or a history of TdP.
   * Have any malignancies or have a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
   * Significant trauma or major surgery within 1 month of the first dose of study drug or considered in imminent need for surgery or with elective surgery scheduled to occur during the study.

   Prior/Concomitant Therapy:
6. Have received any of the prohibited treatment regimens specified.

   Prior/Concurrent Clinical Study Experience:
7. Previous administration with an investigational drug or vaccine that do not affect vitiligo within 4 weeks of Day 1 [Baseline] or within 5 half-lives, whichever is longer.

   Diagnostic Assessments:
8. Any of the following abnormalities in laboratory values at Screening, as assessed by the study-specific laboratory and, if deemed necessary, confirmed by a single repeat:

   * Renal impairment
   * Hepatic dysfunction
9. Screening standard 12-lead ECG that demonstrates clinically relevant abnormalities

   Other Exclusion Criteria:
10. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
11. Adolescent participants 12 to <18 years of age without one of the following:

    * Documented evidence from a health professional of having received varicella vaccination (2 doses); or
    * Evidence of prior exposure to VZV based on serological testing (ie, a positive VZV IgG Ab result) at Screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
US only Co-Primary Endpoints: Response based on Facial Vitiligo Area Scoring Index 75 (F-VASI75) at Week 52 and T-VASI50 at Week 52 | Week 52
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline) and T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
Global (Other than US): Response based on Facial Vitiligo Area Scoring Index 75 (F-VASI75) at Week 52 | Week 52
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline)
Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Adverse Events (AEs), leading to discontinuation, and clinically significant laboratory abnormalities | Baseline through Week 52
  Safety and tolerability of ritlecitinib in participants with nonsegmental vitiligo

SECONDARY OUTCOMES:
US-Only: Response based on F-VASI75 at 24 and 36 weeks | Weeks 24 and 36
  Proportion of participants achieving at least a 75% improvement in F-VASI from Baseline
US-Only: Response based on T-VASI50 at 24 and 36 weeks | Weeks 24 and 36
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
US-Only: Response based on T-VASI75 at 52 weeks | Week 52
  Proportion of participants achieving T-VASI75 (defined as at least 75% improvement in T-VASI from Baseline)
US-Only: Percentage change from baseline (% CFB) in F-VASI at 24, 36, and 52 weeks | Weeks 24, 36, and 52
  Median % CFB in F-VASI in participants treated with ritlecitinib 50 mg QD versus placebo
US-Only: Percentage change from baseline (% CFB) in T-VASI at 24, 36, and 52 weeks | Weeks 24, 36, and 52
  Median % CFB in T-VASI in participants treated with ritlecitinib 50 mg QD versus placebo
US-Only: Patient Global Impression of Severity-Face (PGIS-F) | Week 52
  Proportion of responders based on PGIS-F at 52 weeks
US-Only: Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) | Week 52
  Proportion of responders based on PGIS-V at 52 weeks
Global (Other than US): Response based on F-VASI75 at 24 and 36 weeks | Weeks 24 and 36
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline)
Global (Other Than US): Response based on T-VASI50 at 24, 36, and 52 weeks | Weeks 24, 36, and 52
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
Global (Other than US): Percentage change from baseline (% CFB) in F-VASI at 24, 36, and 52 weeks | Weeks 24, 36, and 52
  Median % CFB in F-VASI in participants treated with ritlecitinib 50 mg QD versus placebo
Global (Other than US): Percentage change from baseline (% CFB) in T-VASI at 24, 36, and 52 weeks | Weeks 24, 36, and 52
  Median % CFB in T-VASI in participants treated with ritlecitinib 50 mg QD versus placebo
Global (Other than US): Patient Global Impression of Severity-Face (PGIS-F) | Weeks 24, 36, and 52
  Proportion of responders based on PGIS-F at 24, 36, and 52 weeks
Global (Other than US): Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) | Weeks 24, 36, and 52
  Proportion of responders based on PGIS-V at 24, 36, and 52 weeks
All Countries: Proportion of participants achieving disease stabilization | Baseline through week 52
  The difference in the proportion of participants with stable disease at all timepoints in participants with non segmental vitiligo treated with ritlecitinib 50 mg QD compared to placebo
Response based on T-VASI50 | Baseline through week 4, week 8, week 12, week 48
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
Response based on F-VASI75 | Baseline through week 4, week 8, week 12, week 48
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline)
Response based on T-VASI75 | Baseline through week 4, week 8, week 12, week 24, week 36, week 48
  Proportion of participants achieving T-VASI75 (defined as at least 75% improvement in T-VASI from Baseline)
Proportion of participants with sustained improvement in T-VASI | Week 36 through week 52
  Defined as maintenance of ≥T-VASI50 from Week 36 to Week 52
Proportion of participants with sustained improvement in F-VASI | Week 36 through week 52
  Defined as maintenance of ≥F-VASI75 from Week 36 to 52
All Countries: Time to rescue medication | Baseline through week 52
  Comparing time to rescue medication curves and difference in probabilities of using rescue medication
Percentage change from baseline in F-VASI | Baseline through week 52
  Median % CFB in F-VASI at appropriate timepoints in participants treated with ritlecitinib 50 mg QD versus placebo
Percentage change from baseline in T-VASI | Baseline through week 52
  Median % CFB in T-VASI at appropriate timepoints in participants treated with ritlecitinib 50 mg QD versus placebo
Response based on T-VASI90 | Baseline through week 52
  Proportion of participants achieving T-VASI90 (defined as at least 90% improvement in T-VASI from Baseline)
Response based on T-VASI100 | Baseline through week 52
  Proportion of participants achieving T-VASI100 (defined as at least 100% improvement in T-VASI from Baseline)
Response based on F-VASI50 | Baseline through week 52
  Proportion of participants achieving F-VASI50 (defined as at least 50% improvement in F-VASI from Baseline).
Response based on F-VASI90 | Baseline through week 52
  Proportion of participants achieving F-VASI90 (defined as at least 50% improvement in F-VASI from Baseline).
Response based on F-VASI100 | Baseline through week 52
  Proportion of participants achieving F-VASI100 (defined as at least 100% improvement in F-VASI from Baseline).
Patient Global Impression of Severity-Face (PGIS-F) | Weeks 24 and 36
  Proportion of responders based on PGIS-F at 24 and 26 weeks
Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) | Weeks 24 and 36
  Proportion of responders based on PGIS-V at 24 and 36 weeks
Patient Global Impression of Change-Face (PGIC-F) | Weeks 24, 36, and 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-F at 24, 36, and 52 weeks
Patient Global Impression of Change- Overall Vitiligo (PGIC-V) | Weeks 24, 36, and 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-V at 24, 36, and 52 weeks
Change from baseline in Dermatology Life Quality Index (DLQI) or Children Dermatology Life Quality Index (CDLQI) | Week 52
  To evaluate the change from baseline in DLQI or CDLQI at week 52
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) | Week 52
  To assess the effect of ritlecitinib compared to placebo on depression and anxiety subscales of the HADS at week 52
The proportion of patients achieving absence of depression on HADS depression subscale | Week 52
  Response based on a 'normal' subscale score indicative of an absence of depression (in participants with baseline HADS subscale scores indicative of depression)
The proportion of patients achieving absence of anxiety on HADS anxiety subscale | Week 52
  Response based on a 'normal' subscale score indicative of an absence of anxiety (in participants with baseline HADS subscale scores indicative of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham Faculty Office Towers (Regulatory, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Marvel Clinical Research, Huntington Beach, California
  - Wallace Medical Group, Inc, Los Angeles, California
  - Audiology, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Center for Dermatology and Dermatologic Surgery, Washington D.C., District of Columbia
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Skin Care Research, Hollywood, Florida
  - Clever Medical Research, Miami, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Olympian Clinical Research, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Advanced Medical Research, PC., Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Velocity Clinical Research at The Dermatology Clinic, Baton Rouge, Baton Rouge, Louisiana
  - DelRicht Research, Baton Rouge, Louisiana
  - The NeuroMedical Center (XRay), Baton Rouge, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Prairieville Family Hospital (XRay), Prairieville, Louisiana
  - Visage Dermatology and Aesthetic Center, Bowie, Maryland
  - Lawrence J Green, MD LLC, Rockville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hamzavi Dermatology - Canton, Canton, Michigan
  - Skin Specialists, PC, Omaha, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Accellacare, Wilmington, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Remington Davis Clinical Research, Columbus, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Alpesh D. Desai, DO PLLC - Research, Houston, Texas
  - Austin Institute for Clinical Research, Houston, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Australia (5):
  - The Skin Hospital, Darlinghurst, New South Wales
  - North Eastern Health Specialists, Campbelltown, South Australia
  - Skin Health Institute Inc., Carlton, Victoria
  - Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Bulgaria (3):
  - MC "Asklepiy" OOD, Dupnitsa
  - DCC Aleksandrovska EOOD, Sofia
  - UMHAT "Prof. dr. Stoyan Kirkovich" AD, Stara Zagora
- Canada (8):
  - Dermatology Research Institute, Calgary, Alberta
  - CaRe Clinic, Red Deer, Alberta
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North York Research Inc, Toronto, Ontario
  - Whitby Health Centre Dermatology trials, Whitby, Ontario
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
  - Centre de Recherche Saint-Louis, Québec
- China (11):
  - Fujian Medical University Affiliated First Hospital, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Hospital of Wuhan, Wuhan, Hubei
  - The First Hospital of China Medical University/Dermatology and STD Department, Shenyang, Liaoning
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital/Dermatology Department, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The first Affiliated hospital of Wenzhou medical University, Wenzhou, Zhejiang
- Germany (4):
  - Praxis Leitz und Kollegen, Stuttgart, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Fachklinik Bad Bentheim, Bad Bentheim, Lower Saxony
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
- Italy (3):
  - Istituto Clinico Humanitas, IRCCS, Rozzano, Milano
  - Istituti Fisioterapici Ospitalieri (IFO), Roma, RM
  - Policlinico S. Orsola- Malpighi, Bologna
- Japan (7):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Sugamo Kobayashi Derma Clinic, Toshima-Ku, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Nippon Medical School Hospital, Tokyo
- Mexico (5):
  - Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
  - Sociedad de Metabolismo Y Corazon Sc, Veracruz
  - Arké SMO S.A de C.V, Veracruz
- Poland (5):
  - DermoDent Centrum Medyczne Aldona Czajkowska Rafał Czajkowski s.c., Osielsko, Kuyavian-Pomeranian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - Dermoklinika - Centrum Medyczne spółka cywilna M. Kierstan, J. Narbutt, A. Lesiak, Lodz, Łódź Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Witokrzyski, Świętokrzyskie Voivodeship
- South Africa (4):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Clinresco Centres, Kempton Park, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - Task Central, Cape Town, Western Cape
- South Korea (4):
  - Dongguk University Ilsan Hospital, Goyang-si, Kyǒnggi-do
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (5):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Clinic de Barcelona, Barcelona
  - AUDIKA, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
- Turkey (Türkiye) (4):
  - Istanbul Universitesi- Cerrahpasa, Cerrahpasa Tip Fakultesi, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Celal Bayar Universitesi Hafta Sultan Hastanesi, Manisa
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981040